CLINICAL TRIAL: NCT06973616
Title: A Prospective Randomized Clinical Trial of Two Types of Aesthetics Crowns Used in Restoration of Carious Primary Molars
Brief Title: A Clinical Trial of Two Types of Aesthetics Crowns for Primary Molars
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 466-2023
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Success Rate
Keywords: Randomized clinical trial; Esthetic crowns; Zirconia crown; Bioflx crown; Primary molars; Deciduous molars

STUDY DESIGN:
Intervention Model Description: A split mouth randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia esthetic crowns (Active Comparator): Zirconia esthetic crowns
  Interventions: Procedure: Zirconia crown
- Bioflx esthetic crowns (Active Comparator): Bioflx esthetic crowns
  Interventions: Procedure: Bioflx crown

INTERVENTIONS:
Procedure: Zirconia crown — A zirconia esthetic crown will be randomly placed on one side of the jaw
  Other Names: Esthetic crown
  Arms: Zirconia esthetic crowns
Procedure: Bioflx crown — A Bioflx esthetic crown will be randomly placed on one side of the jaw
  Other Names: Esthetic crown
  Arms: Bioflx esthetic crowns

SUMMARY:
Currently, prefabricated zirconia crowns have been used as an aesthetic restorative material for primary teeth for a few years. Another recently introduced esthetic crown is the Bioflx™ crown. It is made of a resin polymer and claimed to have high strength , flexibility and durability. The aim of this study is to evaluate and compare the clinical and radiographic success of zirconia crowns to that of Bioflx™ crowns in carious primary molars.

DETAILED DESCRIPTION:
Background: Little is known about aesthetic management of decayed primary posterior teeth in children which often requires full-coverage restorations.

Aim: The aim of this study is to evaluate and compare the clinical and radiographic success of zirconia crowns to that of Bioflx™ crowns in carious primary molars.

Methods: this study design is a split mouth randomized controlled clinical trial including children ages between 4-10 years old. Each patient will receive a zirconia crown and Bioflx™ crown on either side of the maxillary or mandibular arch. Clinical procedure: The patients will be randomly allocated to receive either crown on the first visit, and the other type on the next visit which will be 1-2 weeks after. Children and teeth meeting the inclusion criteria will be included. Crowns will be prepared under local anesthesia and rubber dam isolation. Crowns will be evaluated at 1, 6, 12 and 24-month recall appointments according to pre-set success and failure criteria.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4-10 years
* Healthy child
* Child is cooperative
* Subject has a minimum of two bilateral carious upper or lower primary molars
* Teeth exhibiting carious lesions clinically and radiographically
* Teeth selected should be fully erupted, with no evidence of tooth fracture, and could be isolated adequately for crown cementation

Exclusion Criteria:

* Tooth close to exfoliation
* Medical problems in sbjects
* Children requiring advanced behaviour management
* Those not available for future recalls/ follow up

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinically susccessful | 24 months
  Normal gingiva (no inflammation or edema) Normal occlusion (not high in occlusion) Parent satisfied (as reported) Child satisfied (as reported)

CONTACTS AND LOCATIONS:
Overall Officials: OLA Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holsinger DM, Wells MH, Scarbecz M, Donaldson M. Clinical Evaluation and Parental Satisfaction with Pediatric Zirconia Anterior Crowns. Pediatr Dent. 2016;38(3):192-7. PMID 27306242
- [Result] Donly KJ, Sasa I, Contreras CI, Mendez MJC. Prospective Randomized Clinical Trial of Primary Molar Crowns: 24-Month Results. Pediatr Dent. 2018 Jul 15;40(4):253-258. PMID 30345963
- [Result] Ashima G, Sarabjot KB, Gauba K, Mittal HC. Zirconia crowns for rehabilitation of decayed primary incisors: an esthetic alternative. J Clin Pediatr Dent. 2014 Fall;39(1):18-22. doi: 10.17796/jcpd.39.1.t6725r5566u4330g. PMID 25631720
- [Result] Aiem E, Smail-Faugeron V, Muller-Bolla M. Aesthetic preformed paediatric crowns: systematic review. Int J Paediatr Dent. 2017 Jul;27(4):273-282. doi: 10.1111/ipd.12260. Epub 2016 Aug 17. PMID 27532506